CLINICAL TRIAL: NCT02899325
Title: A Single-blind Study to Evaluate the Efficacy and Safety of 18F-Fluorodeoxygalactose (18F-FDGal) Compared to 18F-Fluorodeoxyglucose (18F-FDG) to Detect Hepatocellular Carcinoma Via PET/CT in Patients With Cirrhosis or Chronic Liver Disease
Brief Title: FDGal PET/CT to Detect Hepatocellular Carcinoma
Status: Withdrawn | Type: Observational
Why Stopped: PIs will not pursue trial due to staff and time constraints
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: H16-01905
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2019-12

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis; Chronic Liver Disease
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Diagnostic PET/CT scans — These PET/CT scans will be performed for diagnostic purposes of hepatocellular carcinoma.
  Other Names: 18F-FDG and 18F-FDGal PET/CT scans

SUMMARY:
Liver cancer is one of the leading causes of cancer death among Asian men. If diagnosed early the disease is treatable with surgery. Current conventional imaging modalities have limitations to early detection. This study proposes to use 18F-FGal and 18F-FDG PET/CT scans to compare the clinical efficacy of diagnosing hepatocellular carcinoma (a type of liver cancer) using these PET/CT scans.

DETAILED DESCRIPTION:
Screening Visit Patients will undergo screening procedures for determining eligibility prior to the first PET/CT examination. For practical reasons and to avoid unnecessary travel for research subjects, the initial screening can be conducted by phone, and completed on the day that the first PET/CT examination is performed. However, the PET/CT scan will only be done for subjects that meet all the eligibility criteria and sign the consent form prior to the examination. All patients should have received the consent form by mail, email or fax, at least 24 hours prior to the screening visit.

Demographics Demographic data including date of birth, gender, height and weight information will be obtained.

Medical History and Concomitant Medications The general medical history up to 3 months of study entry (screening visit) should be recorded at the screening visit. The medical history should include procedural and surgical history within the past year. Cancer history should be recorded on a lifetime basis. Previous medications should be recorded up to 28 days prior to screening visit and up to 1 year for cancer treatment if any. All concomitant medications starting from enrollment of subjects should be recorded on subsequent visits for the PET/CT examinations.

Vital Signs Patient's vital signs will be measured including blood pressure, pulse rate and oxygen saturation, within 60 minutes before and 5-15 minutes after administration of the investigational product at PET/CT visits.

PET/CT Scans Patients who meet all eligibility requirements for entry into the study will undergo both an 18F-FDGal and 18F-FDG PET/CT examinations at the BCCA - Vancouver Centre's Functional Imaging Department. The two scans are to be performed on separate days and must be performed between 1 and 15 calendar days of each other. Each PET/CT scan will require approximately 3 hours of additional time from the subject above standard of care. The screening visit and informed consent, can be performed on the same day as the first PET/CT scan (and before the examination), will take approximately one hour.

Prior to the PET/CT scans, subjects will be instructed to take their usual medications as prescribed by their family physician. Subjects will also be instructed to drink 3 to 4 glasses of water within two hours prior to their scan appointment in order to promote hydration and facilitate urinary clearance of background 18F-FDGal/18F-FDG. Subjects must fast for 6 hours prior to 18F-FDGal and 18F-FDG injection, but can drink water at will.

Upon arrival at the PET Imaging department, all subjects will have their weight recorded prior to 18F-FDGal/18F-FDG injection. A baseline blood pressure, heart rate, and oxygen saturation levels will be recorded within 60 minutes prior to 18F-FDGal/18F-FDG injection, and 5 - 15 minutes after injection.

Each study subject will have an intravenous catheter inserted. The subject will receive a bolus intravenous dose of 18F-FDGal/18F-FDG from the BCCA, at a dose of 237 - 521 MBq for 18F-FDG and 119 - 261 MBq MBq for 18F-FDGal, followed by a 5 - 20 mL normal saline flush. The subject will rest in a comfortable chair for 60 minutes.

Upon completion of the scan, subjects will be free to leave the department and will be encouraged to drink 3-4 extra glasses of water by the end of the day to promote further clearance of the remaining tracer in the urinary tract. Overall, the study will take approximately 3 hours of subject time.

Each patient will be monitored on vital signs, adverse events before and after the intravenously 18F-FDGal/18F-FDG administration. Concomitant medication(s) will also be recorded. All of the 18F-FDGal/18F-FDG PET/CT imaging obtained at all study will be sent to a centralized location in DVD sets for re-labeling purpose to mask the patients' identifiers from readers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 19 years of age.
* Patient who accepts to enter the study by signing written informed consent.
* Patient with performance status ≤ 2 Eastern Cooperative Oncology Group (ECOG).
* Patient with cirrhosis or chronic liver disease suspected to have at least 1 hepatic nodule larger than 1 cm in diameter detected by conventional image (US, CT, MRI).

  * Hepatic nodule is defined as any one of the following conditions: suspicious hepatocellular carcinoma, benign tumor such as hemangioma, adenoma or focal nodular hyperplasia, possible metastatic lesions from other primary malignancy.

Exclusion Criteria:

* Patient has serious allergic history or known allergy to 18F-FDGal or 18F-FDG.
* Patient has received therapy for aforementioned diagnosis before the PET scans
* Patient with known (proven) metastases from a prior malignancy
* Patient has been diagnosed with multiple malignancies.
* Female patient who is pregnant, lactating or planning to become pregnant during the study.
* Patient has participated in other investigational trials within 28 days prior to study enrollment.
* Inability to lie supine for the duration of the imaging studies.
* Subject with active systemic infections, or medical conditions that may significantly affect adequate uptake and elimination of radiotracer.
* Subject with conditions judged by the investigator as unsuitable for the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The purpose of this study is to evaluate the diagnostic utility of 18F-FDGal PET/CT in identifying sites of hepatocellular carcinoma where conventional imaging has not been as effective. Concordance with histology, imaging or follow up will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 18F-FDGal in the diagnosis of HCC on per-patient basis | 6 months
  Determination of sensitivity of both exams when compared with pathology reports (if available) and compared with routine imaging (CT, MRI, US) if available. The treatment group will be declared superior if the lower limit of the 95% two-sided confidence interval of the difference of these two proportions is greater than 0.

SECONDARY OUTCOMES:
Number of participants with 18F-FDGal-related adverse events as assessed by abnormal vital sign measurement | 1 hour
  Vital signs (blood pressure, heart rate and pulse oximetry) will be measured at three time points (before and after injection, and 1 hour after the injection). All values that fall outside of the normal parameters will be assessed by a physician and reported as an adverse event.
Sensitivity of 18F-FDGal in the diagnosis of HCC on per-site basis | 6 months
  Determination of sensitivity of both exams when compared with pathology reports (if available) and compared with routine imaging (CT, MRI, US) if available. The treatment group will be declared superior if the lower limit of the 95% two-sided confidence interval of the difference of these two proportions is greater than 0.
Specificity of 18F-FDGal in the diagnosis of HCC | 6 months
  Specificity of 18F-FDGal and 18F-FDG PET/CT are calculated on per-patient and per-site basis (site=lesion).

CONTACTS AND LOCATIONS:
Overall Officials: Francois Benard, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.